CLINICAL TRIAL: NCT07087639
Title: Safety and Effectiveness Evaluation of Novel MICS Venous Cannula
Brief Title: Novel Venous Cannula Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eurosets S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DE-51-20
Record Dates: First submitted 2025-07-07; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery; Heart Surgery; Cardiopulmonary Bypass; Minimally Invasive Surgical Procedures
Keywords: Venous Cannula; Extracorporeal Circulation; Cardiopulmonary Bypass; Cardiac Surgery; Transfemoral Venous Cannulation; Minimally Invasive Cardiac Surgery (MICS); Medical Device; Pressure Drop; Serious Adverse Events (SAE); Device Safety; Device Performance; Open-label Clinical Trial; Single-arm Study; Monocentric Study; Self-expanding Cannula

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomized, monocentric, one arm clinical investigation with pre-marked medical device
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm - Novel Self-expanding Venous Cannula (Experimental): Participants in this arm will undergo transfemoral venous cannulation using the Novel Self-expanding Venous Cannula during on-pump cardiac surgery procedures. The investigational device is a single-use, sterile polyurethane cannula reinforced with a flexible metallic mesh that allows self-expansion once deployed into the vessel. The device is intended to facilitate efficient venous drainage as part of the extracorporeal circulation system. The study aims to evaluate the device's performance in terms of pressure drop and safety profile.
  Interventions: Device: Self-expanding Venous Cannula

INTERVENTIONS:
Device: Self-expanding Venous Cannula — The intervention consists of a self-expanding venous drainage cannula made of polyurethane and reinforced with a flexible metallic mesh. It is designed for transfemoral insertion during on-pump cardiac surgery, including minimally invasive procedures. Once positioned, the cannula expands to its functional diameter to facilitate efficient blood drainage into the extracorporeal circulation system. The configuration used in this study is 680/730 mm in length, 24 Fr, 3/8" diameter. The device is sterile, single-use, and is inserted once on the day of surgery (Day 0) and removed at the end of the procedure. The cannula is used continuously during cardiopulmonary bypass for a maximum duration of 6 hours and is not reused.

SUMMARY:
This is a prospective, open-label, single-arm, single-center clinical investigation designed to evaluate the safety and performance of a Novel Venous Cannula during on-pump cardiac surgery requiring transfemoral venous cannulation. The investigation aims to assess the pressure drop across the cannula during extracorporeal circulation and the incidence of serious adverse events associated with its use. A total of 42 participants will be enrolled.

DETAILED DESCRIPTION:
This clinical investigation evaluates a Novel Venous Cannula intended for drainage of venous blood during extracorporeal circulation in cardiac surgery. The cannula is made of polyurethane and includes a flexible metallic mesh that allows it to collapse during insertion and expand in situ. It is designed for single use, sterile, and is introduced using a dedicated insertion kit.

The study is a non-randomized, open-label, monocentric, single-arm investigation involving 42 adult patients undergoing elective cardiac surgery requiring transfemoral venous cannulation. The investigation includes three visits: a screening visit (from Day -7 to Day -1), the procedure day (Day 0), and a follow-up visit at Day 7 ± 3 days.

The primary effectiveness outcome is the mean pressure drop (mm Hg) across the cannula required to maintain the target flow rate during surgery. The primary safety outcome is the number of serious adverse events (SAEs) related to the use of the investigational device.

Secondary outcomes include several efficacy-related parameters (e.g., venous line flow, pump flow, cannula positioning, volume of infusion, cardioplegic solution usage, and others), as well as safety outcomes including mortality, cardiovascular events, and neurological complications at 7 days post-procedure.

There is no control group in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent obtained
* Hospitalised patients undergoing transfemoral venous cannulation for on pump cardiac surgery procedure

Exclusion Criteria:

* Active bleeding
* Need of ECLS
* Low platelet count (<150,000)
* Any clinical conditions that contra-indicate the anti-coagulation
* Any clinical condition that, in the opinion of the investigator, may interfere with the procedure
* Subjects participating in any other clinical trial or investigation with a medical device within 3 months before Assessment visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Effectiveness: the mean pressure drop (mm Hg) to maintain the desired flow rate (L/min) during the standard surgical procedure | During the surgical procedure (Day 0)
  Measurement of the mean pressure drop (in millimeters of mercury, mmHg) across the novel venous cannula required to maintain the target blood flow rate (liters per minute) during cardiopulmonary bypass in cardiac surgery patients.
Safety: the number of SAE with the Novel Venous Cannula during the standard surgical procedure | From Day 0 (procedure day) to 7 days post-procedure
  Number of serious adverse events (SAEs) occurring during the surgical procedure that are related or possibly related to the use of the novel venous cannula, including device-related complications, cardiovascular events, and other procedure-associated serious adverse events.

SECONDARY OUTCOMES:
Venous Line Flow During Extracorporeal Circulation Unit of Measure: mL/min | During the surgical procedure (Day 0)
  Measurement of venous line flow during CPB to assess the drainage efficiency of the novel venous cannula.
Mean pump flow during extracorporeal circulation Unit of Measure: L/min/m² | During the surgical procedure (Day 0)
  Mean Pump Flow Indexed to Body Surface Area During CPB
Number of cannulae in the surgical field during surgical procedure Unit of Measure: Count (number) | During the surgical procedure (Day 0)
  Number of Cannulae Positioned in the Surgical Field
Number of cannula tip displacement as detected by TTE/TEE during surgical procedure Unit of Measure: n (%) | During the surgical procedure (Day 0)
  Number of Cannula Tip Displacements Detected by TTE/TEE
Mean increase in free Hb measure during surgical procedure Unit of Measure: mg/dL | During the surgical procedure (Day 0)
  Mean Increase in Free Hemoglobin Levels
Mean volume of infusion during surgical procedure Unit of Measure: mL | During the surgical procedure (Day 0)
  Mean Volume of Infusion Administered
Mean volume of cardioplegic solution Unit of Measure: mL | During the surgical procedure (Day 0)
  Mean Volume of Cardioplegic Solution Administered
Mean speed of aspirators during surgical procedure Unit of Measure: mL/min | During the surgical procedure (Day 0)
  Mean Speed of Aspirators Used
Mean percentage of pump flow increase due to the patient's metabolic needs Unit of Measure: % | During the surgical procedure (Day 0)
  Mean Percentage Increase in Pump Flow Due to Metabolic Needs
Mean volume of recovery blood re-administered during surgical procedure Unit of Measure: mL | During the surgical procedure (Day 0)
  Mean Volume of Recovery Blood Re-Administered
Number of patients for whom blood concentrator was used Unit of Measure: Count (number of patients) | During the surgical procedure (Day 0)
  Number of Patients for Whom a Blood Concentrator Was Used
Presence of echocardiographic abnormalities Unit of Measure: n (%) | During the surgical procedure (Day 0)
  Presence of echocardiographic abnormalities
Number of correctly delivery and deployed Novel Venous Cannula Unit of Measure: Count (number of cannulae) | During the surgical procedure (Day 0)
  Number of Novel Venous Cannulae Correctly Delivered and Deployed
Number of technical success without procedural SAE Unit of Measure: n (%) | During the surgical procedure (Day 0)
  Number of patients in which the device was used successfully without the occurrence of procedural serious adverse events during the procedure.
Number of deaths at 7 days after procedure Unit of Measure: Count (number of patients) | From Day 0 (procedure day) to 7 days post-procedure
  Number of patients who die within 7 days following the surgical procedure involving the use of the novel venous cannula.
Number of cardiovascular deaths at 7 days after procedure Unit of Measure: Count (number of patients) | From Day 0 (procedure day) to 7 days post-procedure
  Number of patients who experience cardiovascular-related death within 7 days following the surgical procedure.
Number of cardiovascular SAEs at 7 days after procedure Unit of Measure: Count (number of patients) | From Day 0 (procedure day) to 7 days post-procedure
  Number of cardiovascular-related serious adverse events (SAEs) occurring within 7 days after the procedure.
Number of stroke at 7 days after procedure Unit of Measure: Count (number of patients) | From Day 0 (procedure day) to 7 days post-procedure
  Number of patients experiencing a clinically confirmed stroke within 7 days following the procedure.
Number minor neurological disorder at 7 days after procedure Unit of Measure: Count (number of patients) | From Day 0 (procedure day) to 7 days post-procedure
  Number of patients experiencing minor neurological disorders within 7 days following the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Cecilia Hospital, Cotignola, RA, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be made available to qualified researchers upon reasonable request to the Sponsor, after study completion and publication of the primary results. Each request will be reviewed on a case-by-case basis in accordance with applicable data protection laws, including the EU General Data Protection Regulation (GDPR) 2016/679, and ethical considerations. Access will be granted through a controlled process to ensure the protection of participant confidentiality.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available starting 6 months after publication of the primary study results, and will remain accessible for 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD) and supporting documents (such as study protocol, statistical analysis plan, and clinical study report) will be available to qualified researchers upon reasonable request.
  Requestors must submit a research proposal describing the intended use of the data. Access will be granted after approval by the Sponsor to ensure compliance with ethical standards and data protection regulations, including GDPR.
  Data will be shared through a secure data-sharing platform or via encrypted transfer under a data use agreement that protects participant confidentiality and limits use to the approved research purposes.
URL: https://www.eurosets.com/it/

REFERENCES:
- [Background] Von Segesser. Venous drainage is key for CPB. The royal Society of Medicine, London. 28th November 2008
- [Background] von Segesser LK, Ferrari E, Delay D, Maunz O, Horisberger J, Tozzi P. Routine use of self-expanding venous cannulas for cardiopulmonary bypass: benefits and pitfalls in 100 consecutive cases. Eur J Cardiothorac Surg. 2008 Sep;34(3):635-40. doi: 10.1016/j.ejcts.2008.05.037. Epub 2008 Jul 16. PMID 18635371
- [Background] Van Praet KM, Kofler M, Meyer A, Sundermann SH, Hommel M, Falk V, Kempfert J. Single-Center Experience With a Self-Expandable Venous Cannula During Minimally Invasive Cardiac Surgery. Innovations (Phila). 2022 Nov-Dec;17(6):491-498. doi: 10.1177/15569845221131534. Epub 2022 Oct 30. PMID 36314445
- [Background] Stoney WS. Evolution of cardiopulmonary bypass. Circulation. 2009 Jun 2;119(21):2844-53. doi: 10.1161/CIRCULATIONAHA.108.830174. No abstract available. PMID 19487602
- [Background] Savini C, Gliozzi G, Martin-Suarez S, Zardin D, Mariani C, Cavalli GG, Folesani G, Pacini D. Femoral Venous Cannulation for Minimally Invasive Surgery: Three Years Experience with Wall-less, Self-expandable Cannula. The International Society for Minimally Invasive Cardiothoracic Surgery 2021, PC110.
- [Background] Pinon M, Pradas G, Molina D, Legarra JJ. Use of self-expanding venous cannula in tricuspid reoperation. Eur J Cardiothorac Surg. 2015 Sep;48(3):499-501. doi: 10.1093/ejcts/ezu492. Epub 2015 Jan 9. PMID 25575788
- [Background] Mueller XM, Mallabiabrena I, Mucciolo G, von Segesser LK. Optimized venous return with a self-expanding cannula: from computational fluid dynamics to clinical application. Interact Cardiovasc Thorac Surg. 2002 Sep;1(1):23-7. doi: 10.1016/s1569-9293(02)00006-3. PMID 17669950
- [Background] Puis L, Milojevic M, Boer C, De Somer FMJJ, Gudbjartsson T, van den Goor J, Jones TJ, Lomivorotov V, Merkle F, Ranucci M, Kunst G, Wahba A; EACTS/EACTA/EBCP Committee Reviewers. 2019 EACTS/EACTA/EBCP guidelines on cardiopulmonary bypass in adult cardiac surgery. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):161-202. doi: 10.1093/icvts/ivz251. No abstract available. PMID 31576402
- [Background] Jegger D, Chassot PG, Bernath MA, Horisberger J, Gersbach P, Tozzi P, Delay D, von Segesser LK. A novel technique using echocardiography to evaluate venous cannula performance perioperatively in CPB cardiac surgery. Eur J Cardiothorac Surg. 2006 Apr;29(4):525-9. doi: 10.1016/j.ejcts.2005.12.050. Epub 2006 Feb 14. PMID 16476552
- [Background] Jegger D, Horisberger J, Boone Y, Seigneuil I, Jachertz M, Holzmann I, von Segesser LK. Vascular access for cardiopulmonary bypass procedures. Artif Organs. 2004 Jul;28(7):649-54. doi: 10.1111/j.1525-1594.2004.07372.x. PMID 15209858
- [Background] Jegger D, Corno AF, Mucciolo A, Mucciolo G, Boone Y, Horisberger J, Seigneul I, Jachertz M, von Segesser LK. A prototype paediatric venous cannula with shape change in situ. Perfusion. 2003 Mar;18(1):61-5. doi: 10.1191/0267659103pf640oa. PMID 12705652
- [Background] Ismail A, Semien G, Sharma S, Collier SA, Miskolczi SY. Cardiopulmonary Bypass. 2024 Aug 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482190/ PMID 29489210
- [Background] Gravlee GP, Davis RF, Kurusz M, Utley JR. Cardiopulmonary Bypass. 2nd Edition. Eugene A, Hessel II, Aaron G. Hill. Chapter 5: circuitry and cannulation - 2016
- [Background] Frederick A, Hensley Jr, Martin DE, Gravlee G. A Practical Approach to Cardiac Anesthesia. 3rd Edition. 2011; Larach DR, Gibbs NM. Chapter 7. Anesthetic Management During Cardiopulmonary Bypass
- [Background] Hessel EA 2nd. A Brief History of Cardiopulmonary Bypass. Semin Cardiothorac Vasc Anesth. 2014 Jun;18(2):87-100. doi: 10.1177/1089253214530045. Epub 2014 Apr 10. PMID 24728884
- [Background] Ceresa F, Mammana LF, Leonardi A, Palermo A, Patane F. Virtually Wall-Less versus Standard Thin-Wall Venous Cannula in the Minimally Invasive Mitral Valve Surgery: Single-Center Experience. Medicina (Kaunas). 2023 Jun 29;59(7):1221. doi: 10.3390/medicina59071221. PMID 37512033
- [Background] Ferrari E, von Segesser LK, Berdajs D, Muller L, Halbe M, Maisano F. Clinical Experience in Minimally Invasive Cardiac Surgery With Virtually Wall-Less Venous Cannulas. Innovations (Phila). 2018 Mar/Apr;13(2):104-107. doi: 10.1097/IMI.0000000000000478. PMID 29677020
- [Background] Abdel-Sayed S, Favre J, Horisberger J, Taub S, Hayoz D, von Segesser LK. New bench test for venous cannula performance assessment. Perfusion. 2007 Nov;22(6):411-6. doi: 10.1177/0267659108089759. PMID 18666745